CLINICAL TRIAL: NCT06910371
Title: Digital Detox Study: A Randomized Controlled Trial
Brief Title: Digital Detox Study
Acronym: RESET
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danube University Krems (Other)
Responsible Party: Principal Investigator, Christoph Pieh, Full Professor, Danube University Krems
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EK GZ 15 2024-2027; EK GZ 15 2024-2027 (Other: University of Continuous Education Krems)
Record Dates: First submitted 2025-03-20; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Prevention; Digital Health; Smartphone Addiction
Keywords: digital detox; screen time reduction; mental health
MeSH Terms: conditions — Internet Addiction Disorder; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with two unblinded parallel groups)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone screen time reduction group (IG) (Experimental): Smartphone screen time reduction group (intervention group = IG) will reduce smartphone screen time for 3 weeks to less-equal than 2 hours. After intervention, there are no screen time predefined values until follow-up.
  Interventions: Behavioral: smartphone screen time reduction
- Control group (No Intervention): Control group (CG) will use smartphone unchanged for 6 consecutive weeks.

INTERVENTIONS:
Behavioral: smartphone screen time reduction — Smartphone screen time has to be reduced to less-equal 2 hours per day for 3 consecutive weeks.
  Arms: Smartphone screen time reduction group (IG)

SUMMARY:
The Digital Detox study is designed as a randomized controlled trial (two unblinded parallel groups) to examine the effects of reducing smartphone screentime on mental health. After giving informed consent, participants will be screened for eligibility. Inclusion criteria are adult subjects (greater-equal 18 years) using their smartphone daily for 3 hours or more, with sufficient German skills and no ongoing psychotherapy, psychological or psychopharmacological treatment. For eligibility screening, participants have to upload a screenshot of their smartphone screen time of the last week, have to state about mental health disorders (self-report) and their sociodemographic variables (age, gender, country of residence, education and professional status, urban/rural nature of place of residence), and have to fill out the following questionnaires: depressive symptoms (PHQ-9), well-being (WHO-5), sleep quality (ISI), stress (PSQ-20), loneliness (three-item loneliness scale), physical activity, and smartphone usage behavior.

If the inclusion criteria are met, participants will be randomized to the intervention or control group. The intervention consists of a three-week screen time reduction to a maximum of 2 hours per day for 3 consecutive weeks. The control group continues to use their smartphones as usual during this time. At the beginning of the study (=baseline T0), all participants will complete the following primary outcome measures (depressive symptoms (PHQ-9), well-being (WHO-5), sleep quality (ISI), stress (PSQ-20)) and secondary outcome measures (loneliness (three-item loneliness scale), craving (CEQ-F), physical activity). Both groups will also complete items on loneliness and physical activity twice during the intervention (after the first and second week of the intervention) to monitor changes in these variables during the intervention. After the three weeks of intervention (post-intervention T1), both groups will again fill out the the same outcome measures as for T0. After the 3-week intervention, there are no further restrictions regarding the participants' smartphone screen time. Follow-up (T2) will be after 3 more weeks and the same outcome measures as for T0 and T1 will be collected.

The weekly smartphone screen time is assessed via self-reporting and screenshot upload. Information is also provided on the weekly activations of the smartphone and a screenshot is uploaded of the most frequently used apps. All data is collected weekly for the previous week.

The study will be performed entirely via a smartphone app (ESMIra), which is designed especially to run longitudinal studies.

Primary hypotheses:

* H1: Reducing smartphone use to a maximum of 2 hours/day over 3 weeks leads to a difference in the depressive symptoms of the intervention participants before and after participating in the intervention.
* H2: Reducing smartphone use to a maximum of 2 hours/day over 3 weeks leads to a difference in the the sleep quality of the intervention participants before and after participating in the intervention.
* H3: Reducing smartphone use to a maximum of 2 hours/day over 3 weeks leads to a difference in perceived stress of the intervention participants before and after participating in the intervention.
* H4: Reducing smartphone use to a maximum of 2 hours/day over 3 weeks leads to a difference in the well-being of the intervention participants before and after participating in the intervention.
* H5: The reduction in smartphone use to a maximum of 2 hours/day over 3 weeks led to a difference in depressive symptoms between the control and intervention groups at the post-intervention time point.
* H6: The reduction in smartphone use to a maximum of 2 hours/day over 3 weeks led to a difference in sleep quality between the control and intervention groups at the post-intervention time point.
* H7: The reduction in smartphone use to a maximum of 2 hours/day over 3 weeks led to a difference in perceived stress between the control and intervention groups at the post-intervention time point.
* H8: The reduction in smartphone use to a maximum of 2 hours/day over 3 weeks led to a difference in well-being between the control and intervention groups at the post-intervention time point.

DETAILED DESCRIPTION:
The study employs a convenience sampling method to recruit participants. Recruitment channels include social media accounts of the university and the department (Instagram: istokay.at, unikrems, and X (formerly Twitter): @PsychiUniKrems), where posts and story updates will provide information about the study. Additionally, emails will be sent to universities, universities of applied sciences, and other educational institutions, and flyers will be distributed. These materials will inform potential participants about the study's purpose and procedures.

Interested individuals can access the study page on ESMira via a link or QR code. There, they provide electronic consent before completing the screening questionnaire, which assesses the study's inclusion and exclusion criteria.

Control group will be offered to also participate in the intervention after study completion.

Data Collection

All data collection and communication with participants will take place exclusively through the ESMira research application. ESMira is compatible with all smartphones and was specifically developed for scientific studies, particularly those with a longitudinal design. The app allows for the administration of questionnaires at pre-specified time points and facilitates fully anonymous communication with participants.

A permanent internet connection is not required for using ESMira. Completed questionnaires are stored locally on the app and automatically uploaded once an internet connection becomes available. Research data is stored in encrypted form on a secure server at the University for Continuing Education Krems. Participant anonymity is ensured through a randomly generated user ID (12 alphanumeric characters, e.g., 4mZm-F8vN-5Vyk) assigned by ESMira.

For more information about ESMira, visit: https://github.com/KL-Psychological-Methodology/.

Data Security and Storage:

In accordance with Article 32 of the DSGVO, data security measures will be implemented to ensure the protection and confidentiality of participant information. The data is stored on a local server and is protected against unauthorized access. Unauthorized reading, copying, modification or deletion is therefore not possible. Furthermore, the data is only collected and stored in pseudonymized form. The personal data is only stored for the duration of the study. After that, it is only stored in a completely anonymized form.

Used questionnaire:

Screening only:

Sociodemographic variables: Age (in years), gender, country of residence, highest completed education, current educational/employment status, urban/rural classification of residence.

Mental health (self-report):

Do you have a mental health condition for which you are currently receiving treatment? (yes/no) Are you currently taking medication for a mental health condition? (yes/no) Smartphone usage: Do you use your smartphone for an average of ≥3 hours per day? (yes/no)

Assessed at screening and all subsequent time points (T0, T1, T2):

Depressive Symptoms (PHQ-9) The Patient Health Questionnaire (PHQ-9) is used to assess depressive symptoms in its validated German version, consisting of 9 items.

Well-being (WHO-5) The validated German version of the World Health Organization Well-Being Index (WHO-5) is used to assess participants' well-being and consists of 5 items.

Sleep Quality (ISI) :

The Insomnia Severity Index (ISI) is used in its validated German version to assess the quality of sleep and consists of 7 items.

Stress (PSQ-20): Stress is assessed using the German version of the short form of the Perceived Stress Questionnaire (PSQ-20), which consists of 20 items.

Loneliness (3-Item Loneliness Questionnaire): Loneliness is assessed using the German version of the Three Items Loneliness Scale, consisting of 3 items.

Physical activity: "On how many of the last 7 days were you physically active for at least 60 minutes?" and "How many minutes did you spend doing sport in the last 7 days?" Craving (CEQ-F) [not in screening]: Craving is measured using the Craving Experience Questionnaire (CEQ-F) in the German version, for behavioral addictions and smartphone use in particular, and consists of 9 items.

Smartphone use (self-report and upload of screenshots of screentime over the last week, activations, and the most frequently used apps).

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects
* greater-equal 18 years
* sufficient German skills
* using a smartphone daily 3 hours or more
* no ongoing psychotherapy, psychological or psychopharmacological treatment

Exclusion Criteria:

* Age under 18 years
* insufficient German skills
* Smartphone use less than 3 hours per day
* ongoing psychotherapy, psychological or psychopharmacological treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2025-05-19 (Estimated); Study Completion 2025-06-09 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms | At baseline (t0), after the intervention period (= three weeks after t0) (t1), and at follow-up (t2) in both groups.
  The Patient Health Questionnaire (PHQ-9) is used to assess depressive symptoms in its validated German version, consisting of 9 items. Higher scores mean a higher level of depressive symptoms.
Well-being | At baseline (t0), after the intervention period (= three weeks after t0) (t1), and at follow-up (t2) in both groups.
  The validated German version of the World Health Organization Well-Being Index (WHO-5) is used to assess participants' well-being and consists of 5 items. Higher scores mean a higher level of well-being.
Sleep quality | At baseline (t0), after the intervention period (= three weeks after t0) (t1), and at follow-up (t2) in both groups.
  The Insomnia Severity Index (ISI) is used in its validated German version.Higher socres mean a higher level of insomnia symptoms.
Stress | At baseline (t0), after the intervention period (= three weeks after t0) (t1), and at follow-up (t2) in both groups.
  Stress will be evaluated with the German version of the 20-item short form of the Perceived Stress Questionnaire (PSQ-20). Higher scores mean a higher level of stress.

OTHER OUTCOMES:
Craving | At baseline (t0), after the intervention period (= three weeks after t0) (t1), and at follow-up (t2) in both groups.
  Craving will be assessed with the validated German version of the Craving Experience Questionnaire (CEQ-F). Higher scores mean a higher level of craving.
Loneliness | At baseline (t0), after the intervention period (= three weeks after t0) (t1), and at follow-up (t2) in both groups.
  Loneliness will be measured with the validated German version of the Three-item-loneliness scale. Higher scores mean a higher level of loneliness.
Physical activity | Weekly from baseline (t0) to post-intervention (t1) (= 3 weeks, 4 times in total), once again at follow-up (t2)
  Self-stated physical activity (times per week as well as minutes per week) will be assessed (self-statement).
Smartphone usage | Weekly from baseline (t0) to follow-up (t2) (= 6 weeks, 7 times in total) in both groups
  Smartphone usage will be assessed weekly in both groups via self-report and screenshot upload regarding the screen time, the activations and the most frequently used apps in the previous weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Pieh, Full Professor, Principal Investigator — University for Continuing Education Krems

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] References: Bastien, C. H., Vallières, A., & Morin, C. M. (2001). Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Medicine, 2(4), 297-307. https://doi.org/10.1016/s1389-9457(00)00065-4 Brandtner, A., & Wegmann, E. (2023). The fear in desire: linking desire thinking and fear of missing out in the social media context. BMC Psychology, 11(1), 176. Brähler, E., Mühlan, H., Albani, C., & Schmidt, S. (2007). Teststatistische Prüfung und Normierung der deutschen Versionen des EUROHIS-QOL Lebensqualität-Index und des WHO-5 Wohlbefindens-Index. Diagnostica, 53(2), 83-96. https://doi.org/10.1026/0012-1924.53.2.83 Cornil, A., Long, J., Rothen, S., Perales, J. C., de Timary, P., & Billieux, J. (2019). The gambling craving experience questionnaire: Psychometric properties of a new scale based on the elaborated intrusion theory of desire. Addictive Behaviors, 95, 110-117. Fliege, H., Rose, M., Arck, P., Walter, O. B., Kocalevent, R.-D., Weber, C., & Klapp, B. F. (2005). The Perceived Stress Questionnaire (PSQ) Reconsidered: Validation and reference values from different clinical and healthy adult samples. Psychosomatic Medicine, 67(1). https://doi.org/10.1097/01.psy.0000151491.80178.78 Fliege, H., Rose, M., Arck, P., Levenstein, S., & Klapp, B. F. (2009). PSQ - Perceived Stress Questionnaire. In. Leibniz Institute for Psychology - Open Test Archive. https://doi.org/https://doi.org/10.23668/psycharchives.5138 Fritz, M. The Craving Experience Questionnaire: Validation of a German Version. Gerber, M., Lang, C., Lemola, S., Colledge, F., Kalak, N., Holsboer-Trachsler, E., Pühse, U., & Brand, S. (2016). Validation of the German version of the Insomnia Severity Index in adolescents, young adults and adult workers: results from three crosssectional studies. BMC Psychiatry, 16, 174. https://doi.org/10.1186/s12888-016-0876-8 Klein, E. M., Zenger, M., Tibubos, A. N., Ernst, M., Reiner, I., Schmalbach, B., ... & Beutel, M. E. (2021). Loneliness and its relation to mental health in the general population: Validation and norm values of a brief measure. Journal of affective disorders reports, 4, 100120. Kroenke, K., Spitzer, R. L., & Williams, J. B. (2001). The PHQ-9: validity of a brief depression severity measure. Journal of General Internal Medicine, 16(9), 606-613. https://doi.org/10.1046/j.1525-1497.2001.016009606.x Levenstein, S., Prantera, C., Varvo, V., Scribano, M. L., Berto, E., Luzi, C., & Andreoli, A. (1993). Development of the perceived stress questionnaire: A new tool for psychosomatic research. Journal of Psychosomatic Research, 37(1), 19-32. https://doi.org/https://doi.org/10.1016/0022-3999(93)90120-5 Löwe, B., Spitzer, R. L., Gräfe, K., Kroenke, K., Quenter, A., Zipfel, S., Buchholz, C., Witte, S., & Herzog, W. (2004). Comparative validity of three screening questionnaires for DSM-IV depressive disorders and physicians' diagnoses. Journal of Affective Disorders, 78(2), 131-140. https://doi.org/10.1016/S0165-0327(02)00237-9 Morin, C. M., Belleville, G., Bélanger, L., & Ivers, H. (2011). The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep, 34(5), 601-608. https://doi.org/10.1093/sleep/34.5.601 Reinwarth, A. C., Petersen, J., Beutel, M. E., Hautzinger, M., & Brähler, E. (2024). Social support in older adults: Validation and norm values of a brief form of the Perceived Social Support Questionnaire (F-SozU K-6). Plos one, 19(3), e0299467. Topp, C. W., Østergaard, S. D., Søndergaard, S., & Bech, P. (2015). The WHO-5 Well- Being Index: A Systematic review of the literature. Psychotherapy and Psychosomatics, 84(3), 167-176. https://doi.org/10.1159/000376585
- See also: This was the first pilot study on the topic, and its results and experiences now serve as the basis for a follow-up study with a significantly larger study sample. The existing literature largely aligns with the findings of this study. — https://bmcmedicine.biomedcentral.com/articles/10.1186/s12916-025-03944-z#Bib1

DOCUMENTS (3):
  • Study Protocol (2025-03-17): https://cdn.clinicaltrials.gov/large-docs/71/NCT06910371/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-19): https://cdn.clinicaltrials.gov/large-docs/71/NCT06910371/SAP_001.pdf
  • Informed Consent Form (2025-03-25): https://cdn.clinicaltrials.gov/large-docs/71/NCT06910371/ICF_002.pdf